CLINICAL TRIAL: NCT00339300
Title: A Case-Referent Study of Brain Tumors in Adults
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999994036; OH94-C-N036
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-02-26

CONDITIONS: Brain Tumors
Keywords: Etiology; Brain Cancer; Epidemiology; Brain Tumors; Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The etiology of brain tumors is poorly understood. Due, in part, to public concern about a postulated relationship between the use of cellular telephones or other increasingly prevalent environmental exposures and the incidence of brain cancer in adults, the National Cancer Institute is collaborating with three U.S. hospitals in a comprehensive case-control study of malignant and benign brain tumors. Factors under consideration include use of cellular phones and other wireless communication devices, workplace exposures to chemical agents and electromagnetic fields, dietary factors, family history of tumors, genetic determinants of susceptibility, home appliance use, reproductive history and hormonal exposures, viruses, medical and dental exposure to ionizing radiation, and other aspects of medical history.

Approximately 800 newly diagnosed brain tumor cases and 800 controls have been enrolled at hospitals in Boston, Phoenix and Pittsburgh. Cases include all adults (age greater than or equal to 18 years) newly diagnosed with a histologically confirmed intracranial glioma, intracranial meningioma or acoustic neuroma. Controls are patients admitted to the same hospitals as the cases, and treated for any of a variety of non-malignant conditions. Participating cases and controls were interviewed in the hospital by a research nurse and asked to complete a self-administered questionnaire and donate a sample of blood. Key features of the study include its large size, the emphasis on rapid ascertainment of incident cases and interview of study subjects rather than surrogate respondents, the use of detailed, job-specific questions developed by industrial hygienists to ascertain occupational exposures, and the storage of blood samples for future evaluation of inherited susceptibility, biomarkers of exposure and gene-environment interactions.

Implementation of the study protocol proceeded without serious problems. There have been no harmful effects on study participants. There have been no complaints from participants or breaches of confidentiality. Continuation of this research involves analysis and reporting of results. As there will be many papers, this process is expected to extend over the next several years.

DETAILED DESCRIPTION:
The etiology of brain tumors is poorly understood. Due, in part, to public concern about a postulated relationship between the use of cellular telephones or other increasingly prevalent environmental exposures and the incidence of brain cancer in adults. The National Cancer Institute is collaborating with three US hospitals in a comprehensive case-control study of malignant and benign brain tumors. Factors under consideration include the use of cellular phones and other wireless communication devices, workplace exposures to chemical agents and electromagnetic fields, dietary factors, family history of tumors, genetic determinants of susceptibility, home appliance use, reproductive history and hormonal exposures, viruses, medical and dental exposures to ionizing radiation, and other aspects of medical history.

Approximately 800 newly diagnosed brain tumor cases and 800 controls have been enrolled at hospitals in Boston, Phoenix, and Pittsburgh. Cases include all adults (age age greater than or equal to 18 years) newly diagnosed with a histologically confirmed intracranial giloma, intracranial meningioma or acoustic neuroma. Controls are patients admitted to the same hospitals as the cases, and treated for any of a variety of non-malignant conditions. Participating cases and controls were interviewed in the hospital by a research nurse and asked to complete a self-administered questionnaire and donate a sample of blood. Key features of the study include its large size, the emphasis on rapid ascertainment of incident cases and interview of study subjects rather than surrogate respondents, the use of detailed, job-specific questions developed by industrial hygienists to ascertain occupational exposures and gene-environment interactions.

Implementation of the study protocol proceeded without serious problems. There have been no harmful effects on study participants. There have been no complaints from participants or breaches of confidentiality. Continuation of this research involves analysis and reporting of results. Numerous publications have resulted from the study and analyses are ongoing.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

Subjects with malignant and benign adult brain tumors from hospitals in Boston, Phoenix and Pittsburgh.

INCLUSION CRITERIA - Controls:

Patients admitted to the same hospitals as the cases, and treated for any of a variety of non-malignant conditions.

EXCLUSION CRITERIA:

Reasons for exclusion of cases included absense of histologic confirmation or ineligible diagnosis (e.g., schwannoma of facial or trigeminal nerve rather than of acoustic nerve).

EXCLUSION CRITERIA - Controls:

Controls were excluded if cancer was responsible for the hospital admission.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1581 (Actual)
Dates: Start 1994-08-19; Study Completion 2018-02-26

PRIMARY OUTCOMES:
Brain Tumor | 07/15/1994

CONTACTS AND LOCATIONS:
Overall Officials: Cari M Kitahara, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Inskip PD, Tarone RE, Hatch EE, Wilcosky TC, Shapiro WR, Selker RG, Fine HA, Black PM, Loeffler JS, Linet MS. Cellular-telephone use and brain tumors. N Engl J Med. 2001 Jan 11;344(2):79-86. doi: 10.1056/NEJM200101113440201. PMID 11150357
- [Background] Brenner AV, Linet MS, Fine HA, Shapiro WR, Selker RG, Black PM, Inskip PD. History of allergies and autoimmune diseases and risk of brain tumors in adults. Int J Cancer. 2002 May 10;99(2):252-9. doi: 10.1002/ijc.10320. PMID 11979441
- [Background] De Roos AJ, Stewart PA, Linet MS, Heineman EF, Dosemeci M, Wilcosky T, Shapiro WR, Selker RG, Fine HA, Black PM, Inskip PD. Occupation and the risk of adult glioma in the United States. Cancer Causes Control. 2003 Mar;14(2):139-50. doi: 10.1023/a:1023053916689. PMID 12749719